CLINICAL TRIAL: NCT02678377
Title: The SLIM Study: Sling and Botox® Injection for Mixed Urinary Incontinence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Friends of Prentice (Other)
Responsible Party: Principal Investigator, Kimberly Kenton, Professor, Departments of Obstetrics and Gynecology, Urology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00201249
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Results first posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: Mixed Urinary Incontinence; Stress Urinary Incontinence; Urgency Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Botulinum Toxins, Type A; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OnabotulinumtoxinA injections (Active Comparator): 100 units of OnabotulinumtoxinA (Botox®) injected into the detrusor (large muscle of the bladder) at the time of sling surgery.
  Interventions: Drug: OnabotulinumtoxinA (Botox ®) Injections
- Saline injections (Sham Comparator): 100 units of saline injected into the detrusor (large muscle of the bladder) at the time of sling surgery.
  Interventions: Drug: Saline Injections

INTERVENTIONS:
Drug: OnabotulinumtoxinA (Botox ®) Injections — OnabotulinumtoxinA (Botox ®) is a neurotoxin, which inhibits acetylcholine release and temporarily relaxes the bladder muscle to inhibit urgency incontinence.
  Other Names: Botox ®
  Arms: OnabotulinumtoxinA injections
Drug: Saline Injections — Saline will be injected into the bladder so that investigators are masked to subject randomization.
  Arms: Saline injections

SUMMARY:
This double-blind randomized controlled trial seeks to find a better treatment for women with mixed urinary incontinence (both stress and urgency incontinence). The primary aim is to determine whether midurethral sling surgery combined with injections of onabotulinumtoxinA (Botox®) into the detrusor muscle of the bladder improves symptoms of mixed urinary incontinence better than sling surgery alone.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing mid-urethral sling surgery
* Have symptoms of both stress and urgency urinary incontinence
* Able to consent, fill out study documents, and complete all study procedures and follow-up visits
* At least 18 years of age
* English speaking
* Be able and willing to learn clean intermittent self catheterization technique

Exclusion Criteria:

* History of recurrent UTI (defined as three culture proven UTIs within last 12 months)
* Systemic neuromuscular disease known to affect the lower urinary tract
* Undergoing concomitant prolapse surgery
* Previous incontinence surgery
* Treatment with anticholinergic medication in the last 2 months
* Previous bladder injection with onabotulinumtoxinA
* Prisoner Status
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-02; Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kenton, M.D., Principal Investigator — Professor, Departments of Obstetrics and Gynecology, Urology
Locations (1):
- Northwestern Medicine Integrated Pelvic Health Clinic, Chicago, Illinois, United States

REFERENCES:
- [Result] Komar A, Bretschneider CE, Mueller MG, Lewicky-Gaupp C, Collins S, Geynisman-Tan J, Tavathia M, Kenton K. Concurrent Retropubic Midurethral Sling and OnabotulinumtoxinA for Mixed Urinary Incontinence: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jan 1;137(1):12-20. doi: 10.1097/AOG.0000000000004198. PMID 33278293

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note: 100 participants were consented and is the enrollment number, but 12 participants cancelled their surgeries after having signed the consent form. Thus, 88 participants were randomized and are included in the analysis.
Period: Overall Study
Arm/Group | OnabotulinumtoxinA Injections | Saline Injections
Started | 45 | 43
Completed | 41 | 37
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Placebo Group/Saline Injections: The placebo arm received intradetrusor saline injections at the time of their sling.
- Onabotulinum Toxin A: The onabotulinum toxin A group received intradetrusor injections of 100 U onabotulinum toxin A and the placebo group received intradetrusor injections of saline at the time of midurethral sling.
- Total: Total of all reporting groups
Arm/Group | Placebo Group/Saline Injections | Onabotulinum Toxin A | Total
Number analyzed (Participants) | 37 | 41 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (10) | 51.1 (10) | 51 (10)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender (only individuals born with female genitalia were included in the study)
  Participants
    Female | 37 | 41 | 78
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 19
  Not Hispanic or Latino | 25 | 27 | 52
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 28 | 32 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 37 | 41 | 78
UDI-6 [Median (Inter-Quartile Range); unit: units on a scale] — Urinary Distress Inventory, Short Form. The scale is (0-100) and higher values indicate a worse outcome.
  units on a scale | 58.3 [54.2 to 75.0] | 66.7 [54.2 to 70.8] | 62.50 [54.17 to 73.96]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Self-reported Mixed Urinary Incontinence Symptoms
Description: Mixed urinary incontinence symptoms will be assessed by the Patient Global Assessment of Improvement (PGI-I) survey, a patient oriented outcome
Time Frame: 3 months after surgery
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Group: The placebo arm received intradetrusor saline injections at the time of their sling.
- Onabotulinim Toxin A Group: Received 100 U intradetrusor onabotulinum toxin A.
Arm/Group | Placebo Group | Onabotulinim Toxin A Group
Number analyzed (Participants) | 37 | 41
Participants | 31 | 34

2. Secondary Outcome: Incontinence Episode Frequency
Description: Incontinence episode frequency will be assessed by a self-report 3-day urinary diary completed by the subject
Time Frame: 3 months after surgery
Population: Incontinence Episode Frequency on 3 day Diary
Measure: Median (Inter-Quartile Range); unit: episodes
Arm/Group | Placebo Group | Onabotulinim Toxin A Group
Number analyzed (Participants) | 37 | 41
episodes | 0 [0 to 2] | 0 [0 to 2]

3. Secondary Outcome: Urinary Incontinence Symptoms and Quality of Life
Description: Urinary incontinence symptoms and quality of life will be assessed by a satisfaction survey completed by the subject. The scale is 0-100. and higher scores indicate worse outcomes.
Time Frame: 3 months after surgery
Population: IIQ-7: Incontinence QOL
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo Group | Onabotulinim Toxin A Group
Number analyzed (Participants) | 37 | 41
units on a scale | 4.8 [0 to 23.8] | 0 [0 to 9.5]

ADVERSE EVENTS:
Time Frame: 3-months
Groups:
- Placebo Group/Saline Injections: Placebo Group/Saline Injections
- Onabotulinum Toxin A Group: 100 U onabotulinum toxin A group
Arm/Group | Placebo Group/Saline Injections | Onabotulinum Toxin A Group
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/37 | 0/41
Other Adverse Events (participants affected / at risk) | 6/37 | 22/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group/Saline Injections (N=37) | Onabotulinum Toxin A Group (N=41)
Reoperation (Renal and urinary disorders) | 1 (1) | 0 (0) — Re-operation for persistent stress incontinence
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group/Saline Injections (N=37) | Onabotulinum Toxin A Group (N=41)
Urinary Retention within 2 Weeks Surgery (Renal and urinary disorders) | 2 (2) | 5 (5)
Urinary Retention between 2 Weeks and 3 Months (Renal and urinary disorders) | 1 (1) | 5 (5)
Mesh Exposure (Renal and urinary disorders) | 1 (1) | 3 (3)
UTI (Renal and urinary disorders) | 2 (2) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT02678377/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT02678377/SAP_001.pdf
  • Informed Consent Form (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT02678377/ICF_002.pdf